CLINICAL TRIAL: NCT00431665
Title: Effect of Elevated Plasma-Free-Fatty-Acids on Renal Hemodynamic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-070699
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2007-02-06 (Estimated); Status verified 2007-02

CONDITIONS: Renal Circulation; Renal Plasma Flow; Glomerular Filtration Rate; Fatty Acids, Nonesterified
Keywords: Renal Plasma Flow; Glomerular Filtration Rate; Free fatty acids
MeSH Terms: interventions — omega-N-Methylarginine; Triglycerides; Heparin; Somatostatin; Insulin; Glucose; Inulin

INTERVENTIONS:
Drug: NG-monomethyl-L-Arginine (L-NMMA)
Drug: triglycerides (Intralipid 20%)
Drug: heparin
Drug: somatostatin
Drug: insulin
Drug: glucose
Drug: inulin
Drug: paraamino hippurate (PAH)

SUMMARY:
Type 2 diabetes is frequently associated with elevation of plasma-free fatty acids (FFA). Studies indicate that elevation of plasma-FFA induces insulin resistance and also causes endothelial dysfunction as well as hemodynamic changes which are supposed to be involved in the pathogenesis of diabetic vascular disorders.

Glomerular hyperfiltration, which is associated with glomerular hypertension and hypertrophy, a common finding in the early course of type 1 diabetes as well as type 2 diabetes, plays an important role in the development and progression of diabetic nephropathy. These hemodynamic changes are not well understood, but are most likely induced by dilatation of the (precapillary) glomerular arteriole.

In humans the hemodynamic effect of FFAs has so far been investigated locally in brachial and femoral arteries and recently in the eye and skin, where FFAs induced a pronounced increase in blood flow probably due to a local decrease in vascular resistance.

The aim of the present study is to characterise the hemodynamic effects of FFAs in the kidney. In addition we want to test the hypothesis that FFA-induced changes are mediated via endothelial derived nitric oxide (NO). The results of this study could provide information to what extent elevated FFA-plasma levels contribute to hyperfiltration in the early course of diabetes mellitus. The measurements will be done at baseline and during 4 hour infusion of a triglyceride or placebo infusion, combined with heparin.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years
* Body mass index between 15th and 85th percentile (Must et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Evidence of hypertension, pathologic hyperglycemia, hyperlipidemia
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9
Dates: Start 1999-07; Study Completion 2000-06

PRIMARY OUTCOMES:
Renal plasma flow
Glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, MD, Principal Investigator — Department of Internal Medicine III, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria